CLINICAL TRIAL: NCT03603028
Title: Mixed Reality Gaming for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: From The Future LLC (Unknown)
Responsible Party: Principal Investigator, David A Brown, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F89635687
Record Dates: First submitted 2018-04-30; First posted 2018-07-27 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Low Back Pain
Keywords: Walking; Exercise; Exergaming
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exergaming (Experimental)
  Interventions: Device: Exergaming

INTERVENTIONS:
Device: Exergaming — Mixed Reality Gaming for Chronic Low Back Pain
  Other Names: Mixed Reality

SUMMARY:
Mixed Reality Gaming for Chronic Low Back Pain

DETAILED DESCRIPTION:
The company, From the Future and University of Alabama at Birmingham (UAB) team aimed to develop a virtual reality (VR) game that integrated with the features of a specialized self-driven treadmill to provide accessible and progressive walking challenges for individuals with chronic low back pain (LBP). The game was designed to go beyond typical VR research efforts and provide a truly immersive and engaging experience that would motivate individuals with high pain-related fear to keep moving.

ELIGIBILITY:
Inclusion Criteria:

History of chronic low back pain

Exclusion Criteria:

No major neurological, cardiac, pulmonary, or other orthopedic injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Brown, PT, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One individual was unable to participate in Days 2, 3, and followup of the protocol.
Period: Overall Study
Arm/Group | Exergaming
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One participant withdrew from the study
Arm/Group | Exergaming
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Walking Distance
Description: How far participants walk while playing the game as measured by a meter on the instrumented treadmill.
Time Frame: Day 1 through Day 3 of study
Population: One participant withdrew from the study
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Exergaming
Number analyzed (Participants) | 12
meters | 1,134.24 (200.14)

2. Secondary Outcome: Walking Speed
Description: How fast participants walk while playing the game by dividing the distance people walked by the amount of time that they walked
Time Frame: Day 1 - Day 3 of study
Population: One participant withdrew from the study
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Exergaming
Number analyzed (Participants) | 12
meters per second | 1.05 (0.19)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Exergaming
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03603028/Prot_000.pdf